CLINICAL TRIAL: NCT05177380
Title: Efficacy of a Personalized Rehabilitation Program of Facial Involvement in Systemic Sclerosis
Acronym: PREVISS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8072; 2020-A03314-35 (Other: IDRCB)
Record Dates: First submitted 2021-11-22; First posted 2022-01-04 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Systemic Sclerosis; Face; Facial Involvement; Rehabilitation
Keywords: Face; Facial involvement; Rehabilitation; Systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized rehabilitation program of facial involvement in systemic sclerosis (Experimental): 3 sessions of 2 hours of facial rehabilitation in hospital over 2 weeks including:
  * Physiotherapy with facial and endo-oral massages, self-massages, active and passive exercises of the face and mouth, tongue exercises
  * Speech therapy with mobilization of the orofacial sphere applied to swallowing and speech difficulties
  * Individual workshop on the theme of dry mouth, dry mouth, swallowing disorders, and oral care
  * Individual therapeutic makeup workshop
  * A motivational interview
  * A patient notebook with a personalized protocol for self-rehabilitation of the face
  * A video tutorial for self-rehabilitation of the face Facial self-rehabilitation sessions at home
  Interventions: Procedure: Personalized rehabilitation program of facial involvement in systemic sclerosis
- Routine care (Other): Delivery of a standard prescription for facial rehabilitation
  Interventions: Other: Delivery of a standard prescription for facial rehabilitation

INTERVENTIONS:
Procedure: Personalized rehabilitation program of facial involvement in systemic sclerosis — Personalized rehabilitation program of facial involvement in systemic sclerosis
  Arms: Personalized rehabilitation program of facial involvement in systemic sclerosis
Other: Delivery of a standard prescription for facial rehabilitation — Delivery of a standard prescription for facial rehabilitation
  Arms: Routine care

SUMMARY:
Systemic sclerosis is a rare autoimmune disorder characterized by microangiopathy, activation of the immune system, and sclerosis of tissues including the skin. Facial involvement is frequent and disabling. It causes significant functional and aesthetic discomfort, and a major deterioration in quality of life. It results in a loss of suppleness of the skin and subcutaneous tissues, dysfunction of the temporomandibular joint, peribuccal rhagades, microstomia, and dry mouth causing difficulties in mouth opening, feeding, dental care, and weight loss.

Facial involvement in systemic sclerosis can be assessed using the Mouth Handicap in Systemic Sclerosis (MHISS) score, a validated patient questionnaire assessing the functional and aesthetic consequences of systemic sclerosis on the face.

Although common and disabling, facial involvement is underestimated and poorly managed. Immunosuppressive and/or anti-fibrosis drugs are not very effective. Facial rehabilitation could significantly improve the mouth handicap but facial rehabilitation is not currently performed in standard care in systemic sclerosis patients.

The aim of the study is to evaluate the efficacy of a personalized rehabilitation program vs standard care in facial involvement of systemic sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yo
* Systemic sclerosis according to the 2013 ACR/EULAR (American College of Rheumatology) classification criteria
* Systemic sclerosis with facial involvement defined by a MHISS score > 6
* Immunosuppressive and/or anti-fibrosis treatment stable for at least 1 month
* Subject able to understand the objectives and risks of research and to give informed consent
* Subject enrolment in the health insurance scheme

Exclusion Criteria:

* Pregnancy
* Previous participation in a rehabilitation program of facial involvement
* Patient under legal protection
* Impossibility to give clear information of subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Mouth Handicap In Systemic Sclerosis (MHISS) score | Week 6
  A 12-item questionnaire specifically quantifying mouth disability in systemic sclerosis

SECONDARY OUTCOMES:
Mouth Handicap In Systemic Sclerosis (MHISS) score | Week 2
  A 12-item questionnaire specifically quantifying mouth disability in systemic sclerosis
Mouth Handicap In Systemic Sclerosis (MHISS) score | Week12
  A 12-item questionnaire specifically quantifying mouth disability in systemic sclerosis
Interincisal distance measurement | Week 6
  Interincisal distance measurement in mm
Interincisal distance measurement | Week 12
  Interincisal distance measurement in mm
Rodnan skin score on the face | Week 6
  a measure of skin thickness
Rodnan skin score on the face | Week 12
  a measure of skin thickness
Visual Analog Scale (VAS) for pain | Week 2
Visual Analog Scale (VAS) for pain | Week 6
Visual Analog Scale (VAS) for pain | Week12
HAQ questionnaire | Week 6
  Health Assessment Questionnaire
HAQ questionnaire | Week 12
  Health Assessment Questionnaire
SF12 questionnaire (12-item Short Form Survey) | Week 6
  a 12-item general health questionnaire
SF12 questionnaire (12-item Short Form Survey) | Week 12
  a 12-item general health questionnaire
Weight | Week 12
  Weight in kg
Total number of rehabilitation sessions | Week 6
Total duration of rehabilitation sessions | Week 6
Total number of rehabilitation sessions | Week 12
Total duration of rehabilitation sessions | Week 12